CLINICAL TRIAL: NCT05684705
Title: A Single Center, Open-label Study to Investigate the Penetration of Rifabutin Into the Lung After Multiple Intravenous Administrations of BV100 (rifabutin for Infusion) in Healthy Participants
Brief Title: Study to Investigate the Penetration of Rifabutin Into the Lung After Multiple Intravenous Administrations of BV100
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: BioVersys AG (Industry)
Collaborators: CW-Research and Management GmbH (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BV100-004
Record Dates: First submitted 2023-01-05; First posted 2023-01-13 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2024-08

CONDITIONS: Bacterial Infections
MeSH Terms: conditions — Bacterial Infections | interventions — Rifabutin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- BV100 (Experimental): 7 doses of BV100 (q12h)
  Interventions: Drug: BV100

INTERVENTIONS:
Drug: BV100 — Intravenous infusion
  Other Names: Rifabutin for Infusion

SUMMARY:
Study to Investigate the Penetration of Rifabutin Into the Lung After Multiple Intravenous Administrations of BV100

DETAILED DESCRIPTION:
This is a single center, open-label, monocentric, multiple IV dose, phase I study to investigate the penetration of rifabutin into the lung after multiple intravenous administrations of BV100 (rifabutin for infusion) in healthy participants.

ELIGIBILITY:
Inclusion Criteria:

1. Participants who can understand and follow instructions during the study.
2. Participants have been informed both verbally and in writing about the objectives of the clinical trial, the methods, the potential risks, and the discomfort to which he/she may be exposed and has given written consent to participation in the trial prior to trial start and any trial-related procedure.
3. Healthy male participants ≥ 18 and ≤ 55 years of age, or female participants ≥ 18 and ≤ 55 years of age of non-childbearing potential defined as follows:

   * Female participants 50 years of age or older, in menopause for 24 consecutive months and not receiving any hormone replacement therapy within 24 months prior to inclusion into the study
   * female participants who underwent surgical sterilization
   * female participants who underwent hysterectomy
   * female participants with documented premature ovarian failure
4. Healthy participants as defined by absence of evidence of any active or chronic disease following a detailed medical and surgical history, 12-lead ECG, vital signs, physical examination, spirometry (FEV1 > 75% of predicted), and clinical laboratory tests.
5. Weight within a BMI range of 19.0 30.0 kg/m2 inclusive.
6. Healthy male participants with female partners of child-bearing potential must use two methods of contraception, one of which must be a barrier method (e.g., condom) to be used for the duration of the study and for 8 weeks after last IMP dose.
7. Non-smokers, i.e., one who has abstained from use of tobacco or other nicotine containing products for at least 12 months, confirmed by negative cotinine test.
8. Having had no febrile or significant infectious illness for at least one month prior to dosing.
9. The subject is available to complete the study.
10. The subject is able and willing to comply with the restrictions and requirements of the protocol and, in the opinion of the study physician, can complete the study.

Exclusion Criteria:

1. As a result of the medical screening process, the study physician considered the subject unfit for the study.
2. Pregnant or lactating women, or men with female partners, who are not willing to use contraception as defined in inclusion criterion #6.
3. Known or suspected history of hypersensitivity to rifabutin or excipients or to drugs of a similar chemical class including rifampicin, rifapentine, rifaximin; history of allergic reactions leading to hospitalization or any other allergic conditions (including drug allergies, asthma, eczema, anaphylactic reactions but excluding untreated, asymptomatic, seasonal allergies) which the investigator considers may affect the safety of the subject and/or outcome of the study.
4. History of antibiotic associated severe diarrhea within the last year.
5. Any medication that inhibits tubular secretion (e.g., Probenecid, H2 receptor antagonists, trimethoprim) within 2 weeks prior to first dosing.
6. Participants with ECG abnormalities (history, or evidence of second-degree heart block of Mobitz type II, third degree heart block, or any abnormality considered relevant by the investigator), QTcF > 450 ms, PR > 210 ms, or QRS duration > 120 ms.
7. Supine systolic blood pressure > 140 mm Hg or < 90 mm Hg or diastolic blood pressure > 90 mm Hg or < 45 mm Hg at Screening or Day 1 prior to dosing (any abnormal blood pressure results may be repeated once and if the repeat result is within the normal range, it is not considered to have met the exclusion criterion). Pulse rate> 90 bpm or < 45 bpm at Screening.
8. Clinically relevant abnormal values for leukocytes (total WBC), neutrophils, and lymphocytes (total), or values below the lower limit of normal (LLN) at screening. Any abnormal value of these parameters may be repeated and if the repeat result is within the laboratory reference range or not considered relevant by the investigator, it is not considered to have met the exclusion criterion.
9. Alanine aminotransferase (ALT), aspartate aminotransferase (AST), alkaline phosphatase (ALP) and creatinine, above the ULN at Screening. Any abnormal value of these parameters may be repeated and if the repeat result is within the laboratory reference range, it is not considered to have met the exclusion criterion.
10. Any clinical laboratory deviation that is assessed as clinically significant by the investigator (Note the exceptions mentioned in Ex 8 and 9)
11. History of symptomatic, chronic or recurrent infection (e.g., nausea, vomiting, diarrhea, infection with fever) or any viral (including symptomatic herpes zoster), bacterial (including upper respiratory infection), fungal (non-cutaneous) or parasitic infection within 30 days prior to admission to the clinical unit.
12. A positive pre-study serology test for hepatitis B surface antigen (HbsAg), hepatitis C virus (HCV) antibodies or human immunodeficiency virus (HIV)-1 and/or 2 antibodies.
13. A positive drug/alcohol screen at screening or day -1.
14. History of epilepsy, seizures, other neurological disorders, or neuropsychiatric conditions.
15. Participants who have received any prescribed systemic or topical medication within 2 weeks of the first dose administration or five times the elimination half-life (whichever is longer).
16. Participants who had used any non-prescribed systemic or topical medication (including herbal remedies) or megadose vitamins (i.e., 20 to 600 times the recommended daily supplement dose) within 7 days prior to dosing, unless in the opinion of the study physician the medication did not interfere with the study procedures or compromise safety.
17. Participants who have received any medications, including St John's Wort, known to chronically alter drug absorption or elimination processes within 14 days of the first dose administration.
18. Regular use of any inducer of metabolism (e.g., barbiturates, rifampin), or medications interfering with Cytochrome P450, Family 3, Subfamily A (CYP3A) are prohibited, comprising inducers, substrates, and inhibitors in the 3 months prior to the first admission to the clinical unit.
19. Any medication that inhibits active tubular secretion (e.g. Probenecid, H2 receptor antagonists, trimethoprim) within 2 weeks prior to first dosing.
20. Participants who have participated in a clinical study involving administration of an investigational drug (new chemical entity) within the following time-period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
21. Participants who consume more than 21 units of alcohol per week or who have a significant history of alcoholism or drug/chemical abuse (one unit of alcohol equals 285 mL of beer [½ pint], one glass [125 mL] of wine, or 30 mL of 40% alcohol by volume distilled spirits).
22. Excessive consumption of caffeine- or xanthine-containing food or beverages (> 5 cups of coffee a day or equivalent) or inability to stop consuming from 48 hours prior to administration of study treatment.
23. Any use of drugs-of-abuse or alcohol abuse within 2 years prior to the first admission to the clinical unit.
24. Inability to understand or communicate reliably with the investigator or considered by the investigator to be unable to or unlikely to co-operate with the requirements of the study.
25. Any other conditions or factors which in the opinion of the investigator may interfere with study conduct. Failure to satisfy the investigator of fitness to participate for any other reason.
26. Any significant blood loss: donated one unit (450 mL) of blood or more or received a transfusion of any blood or blood products within 60 days, or donated plasma within 7 days prior to the first admission to the clinical unit.
27. Participants who are study site employees or immediate family members of the study site or sponsor employees.
28. Suspected SARS CoV 2 infection

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-10-30 (Actual); Study Completion 2024-12-30 (Actual)

PRIMARY OUTCOMES:
To assess plasma concentration of rifabutin in healthy participants | 5 Days
  Plasma concentration of rifabutin
To assess epithelial lining fluid concentration of rifabutin in healthy participants | 5 days
  Concentration of rifabutin in the epithelial lining fluid
To assess concentration of rifabutin in alveolar macrophages of healthy participants | 5 days
  Concentration of rifabutin in the alveolar macrophages

SECONDARY OUTCOMES:
Safety and Tolerability of multiple dose administration of BV100 in healthy participants | 13 days
  Number of Participants with Treatment-Emergent Adverse Events

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Husband, MD, Study Director — BioVersys SAS
Locations (1):
- Medical University of Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No